CLINICAL TRIAL: NCT04645888
Title: Evaluation of the Effects of Articaine and Bupivacaine in Impacted Third Molar Tooth Surgery
Brief Title: Articaine and Bupivacaine in Impacted Tooth Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Fatih Mehmet Coskunses, Associate Proffesor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 1
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Intervention Model Description: Randomized, split-mouth, triple-blinded study was designed.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This was a triple-blinded study in which the surgeon, the patient and the statistician who performed the data analysis did not know which anesthetic solution had been used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Articaine (Active Comparator): All surgeries were performed by the same surgeon and monitored by the same person. 4 % articaine with 1:200.000 epinephrine was administered to the patients in regional block of the inferior alveolar nerve technique at the first surgery. At the second intervention, patients received the other anesthetic solution which was not used at the first intervention.
  1.5 cc of the solution was used to anesthetize the inferior alveolar and lingual nerve and the remaining 0.5 cc was infiltrated to anesthetize the buccal nerve.
  Interventions: Procedure: Impacted tooth surgery
- Bupivacaine (Active Comparator): All surgeries were performed by the same surgeon and monitored by the same person. % 0.5 bupivacaine without epinephrine was administered to the patients in regional block of the inferior alveolar nerve technique at the first surgery. At the second intervention, patients received the other anesthetic solution which was not used at the first intervention.
  1.5 cc of the solution was used to anesthetize the inferior alveolar and lingual nerve and the remaining 0.5 cc was infiltrated to anesthetize the buccal nerve.
  Interventions: Procedure: Impacted tooth surgery

INTERVENTIONS:
Procedure: Impacted tooth surgery — Surgical extraction of İmpacted tooth

SUMMARY:
Articaine is a common local anesthetic used in oral surgery and belongs to the amide group of it has fast onset with little side effects. Bupivacaine is preferred in prolonged surgical procedures with its long duration of action and residual analgesic effect.

The aim of this study was to evaluate the anesthetic, analgesic, hemodynamic effects of 4% articaine and 0.5% bupivacaine in extraction of impacted mandibular third molar teeth in intraoperative and postoperative periods. Hemodynamic parameters, onset of anesthetic action, total amount, intraoperative comfort, intraoperative bleeding, duration of postoperative anesthesia and analgesia, rescue analgesic use, maximum incisal opening and postoperative pain at 6th, 12th, 24th, 48th and 72th hours and 7th day using a visual analogue scale be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age with bilaterally symmetric, impacted or partially impacted mandibular third molar and patients classified in American Society of Anesthesiologists (ASA) 1 group.

Exclusion Criteria:

* Patients with the presence of any systemic diseases, patients allergic to articaine and bupivacaine or any other NSAIDs and patients with analgesic or anti-inflammatory drugs usage in 15 days before to the surgery.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Changes | 60 minutes
  Systolic and diastolic blood pressure, cardiac rate and blood oxygen saturation level were monitored using a patient monitor before beginning of the surgery (T1), 1 min later following the anesthesia (T2) and immediately after the surgery (T3).
Postoperative pain | 1 week
  Postoperative pain was evaluated by Visual Analogue Scale (VAS) ranging from 0 to 10 and patients were instructed to complete the scale in 6th, 12th, 24th, 48th and 72th hours and 7th day postoperatively.

SECONDARY OUTCOMES:
Maximum mouth opening | 7days
  Maximal incisal opening (MIO) measured with ruler preoperatively and at the 7th day.
Duration of Surgery | 60 minutes
  Duration of the surgery, which was determined by the time between the first incision to last suture was recorded.
Onset of anesthetic action | 10 minutes
  Onset of anesthetic action was be determined by the first sign of numbness of the ipsilateral lower lip, tongue and alveolar mucosa,
Operation time | 60 minutes
  The time between the first incision and the last suture was evaluated as operation time.
Quality of the anesthesia | 60 minutes
  The quality of the anesthesia was evaluated by the surgeon which was based on a 3- point category rating scale: Grade 1: no discomfort reported by the patient during the surgery; Grade 2: any discomfort reported by patient during the surgery, without the need of additional anesthesia; Grade 3: any discomfort reported by patient during the surgery, with the need of additional anesthesia.
Intraoperative bleeding | 60 minutes
  Intraoperative bleeding was rated by the surgeon which based on a 3-point category rating scale as: Grade 1: minimal bleeding; Grade 2: normal bleeding; Grade 3: excessive bleeding.
Surgical difficulty | 60 minutes
  Surgical difficulty was determined by modified Parant scale as follows:
  Grade 1: extraction with forceps only; Grade 2: extraction by osteotomy; Grade 3: extraction by osteotomy and coronal section; Grade 4: complex procedures (root section).
Duration of the postoperative anesthesia | 6 hours
  Duration of the postoperative anesthesia be determined by the absence of sensibility of ipsilateral lower lip, tongue and alveolar mucosa and duration of the postoperative analgesia determined by the time from the end of the operation to the first naproxen sodium intake.

CONTACTS AND LOCATIONS:
Overall Officials: Berkay Tokuc, DDS, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University Faculty of Dentistry, Kocaeli, Basiskele, Turkey (Türkiye)